CLINICAL TRIAL: NCT00356252
Title: Functional Bioavailability of Carotenoids in Humans
Brief Title: Biological Functions of Carotenoids in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: BASF (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: HNRCA1860; PV1087
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Oxidative DNA Damage

INTERVENTIONS:
Drug: mixed carotenoids

SUMMARY:
This study will examine the the efficiency fo absorption of major plant pigments, carotenoids, (lutein, beta-carotene and lycopene)and will measure the biological functions of carotenoids in healthy women in response to an 8-week period of carotenoid supplementation.

The antioxidant capacity (in both the aqueous and lipid compartments), DNA oxidation (single cell gel electrophoresis), Insulin-like Growth Factor (IGF-1), Insulin-like Growth Factor Binding Protein-3 (IGFBP-3), (gene expression profile (high-density filter-based cDNA microarrays), lipid peroxidation (MDA analysis and Isoprostane determination), and antioxidant nutrient levels (carotenoids, tocopherols, ascorbic acid and uric acid) in the circulation will be measured every other week throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* normal hematologic parameters, normal serum albumin, normal liver function, normal kidney function, absence of fat malabsorption and no drug intake which would interfere with fat absorption, metabolism or blood clotting.

Exclusion Criteria:

* Subjects with a history of kidney stones, active small bowel disease or resection, atrophic gastritis, hyperlipidemia, insulin-requiring diabetes, alcoholism, pancreatic disease, or bleeding disorders. Exogenous hormone users, smokers. Subjects weighing greater than 20% above or below the NHANES median standard.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-04; Study Completion 2003-12

PRIMARY OUTCOMES:
DNA damage
plasma carotenoid concentrations

SECONDARY OUTCOMES:
lipid peroxidation
Total antioxidant capacity

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Jin Yeum, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA-Human Nutrition Research Center on Aging, Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Result] Zhao X, Aldini G, Johnson EJ, Rasmussen H, Kraemer K, Woolf H, Musaeus N, Krinsky NI, Russell RM, Yeum KJ. Modification of lymphocyte DNA damage by carotenoid supplementation in postmenopausal women. Am J Clin Nutr. 2006 Jan;83(1):163-9. doi: 10.1093/ajcn/83.1.163. PMID 16400064
- See also: Article — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=PubMed&dopt=Citation&list_uids=16400064